CLINICAL TRIAL: NCT06251024
Title: A Phase IIb, Randomized, Placebo-controlled Study to Evaluate the Efficacy, Safety, and Immunogenicity of an RSV Vaccine Candidate in Adult Participants 60 Years and Older
Brief Title: Study of a Respiratory Syncytial Virus Candidate Formulation in Adults Aged 60 Years and Older
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAE00017; U1111-1271-1514 (Other: ICTRP); VAE00017 (Other: Sanofi Identifier)
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Respiratory Syncytial Virus Infection; Healthy Volunteers
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Intervention Model Description: Parallel, multi-center, case driven
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: * Investigators, laboratory personnel, sponsor and participants will be blinded
  * Study staff preparing/administering the study interventions will be unblinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: RSV vaccine candidate (Experimental): Participants will be enrolled in a 1:1 ratio to receive a single IM administration of the RSV vaccine candidate.
  Interventions: Biological: RSV vaccine candidate
- Group 2: placebo (Placebo Comparator): Participants will be enrolled in a 1:1 ratio to receive a single IM administration of the placebo.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: RSV vaccine candidate — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular Injection
  Arms: Group 1: RSV vaccine candidate
Biological: Placebo — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular Injection
  Arms: Group 2: placebo

SUMMARY:
The purpose of this Phase IIb study is to evaluate the efficacy of the RSV vaccine candidate for the prevention of lower respiratory tract disease (LRTD) due to RSV.

The study will enroll approximately 4500 adults aged 60 years and older in a 1:1 ratio to receive a single intra-muscular (IM) administration of either a pre-determined dose of the RSV vaccine candidate or placebo.

DETAILED DESCRIPTION:
Study duration per participant:

6 months.

Treatment Duration:

1 IM injection. Participants will be followed for approximately 6 months post- vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years or older on the day of inclusion
* A female participant is eligible to participate if she is not pregnant or breastfeeding and:

  • Is of non-childbearing potential. To be considered of non-childbearing potential, a female must be postmenopausal for at least 1 year or surgically sterile.
* Participants with high-risk medical conditions who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion.

Exclusion Criteria: Participants are excluded from the study if any of the following criteria apply:

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known systemic hypersensitivity to any of the study intervention components (eg, polyethylene glycol, polysorbate); history of a life-threatening reaction to the study interventions used in the study or to a product containing any of the same substances ;any allergic reaction (eg, anaphylaxis) after administration of an mRNA vaccine
* History of RSV-associated illness, diagnosed clinically, serologically, or microbiologically in the last 12 months
* Previous history of myocarditis, pericarditis, and/or myopericarditis
* Thrombocytopenia, contraindicating IM injection based on investigator's judgment
* Bleeding disorder or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM injection
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with study conduct or completion
* Alcohol, prescription drug, or substance abuse that, in the opinion of the investigator, might interfere with the study conduct or completion
* Receipt of any vaccine in the 4 weeks preceding any study intervention administration or planned receipt of any vaccine in the 4 weeks following any study intervention administration
* Receipt of any mRNA vaccine in the 60 days preceding any study intervention administration or planned receipt of any mRNA vaccine in the 60 days following any study intervention administration
* Previous vaccination against RSV with a licensed or investigational vaccine or planned receipt during study participation, of vaccination against RSV with a licensed or investigational vaccine other than the study vaccine
* Receipt of immune globulins, blood, or blood-derived products in the past 3 months
* Participation at the time of study enrollment (or in the 4 weeks preceding the first study intervention administration) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure Note: The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4541 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-03-11 (Actual)

PRIMARY OUTCOMES:
Presence of the first episode of RSV-LRTD (RSV A and/or RSV B) ≥ 14 days after vaccination | ≥ 14 days after vaccination
  Number of participants experiencing RSV-LRTD (RSV A and/or RSV B) ≥ 14 days after vaccination

SECONDARY OUTCOMES:
Presence of the first episode of RSV-ARD (RSV A and/or RSV B) ≥ 14 days after vaccination | ≥ 14 days after vaccination
  Number of participants experiencing RSV-ARD (RSV A and/or RSV B) ≥ 14 days after vaccination
Presence of the first episode of RSV MAARD (RSV A and/or RSV B) ≥ 14 days after vaccination | ≥ 14 days after vaccination
  Number of participants experiencing RSV-MAARD (RSV A and/or RSV B) ≥ 14 days after vaccination
Presence of the first episode of RSV LRTD (RSV A) occurring ≥ 14 days after vaccination) | ≥ 14 days after vaccination
  Number of participants experiencing RSV-LRTD (RSV A) ≥ 14 days after vaccination
Presence of the first episode of RSV LRTD (RSV B) occurring ≥ 14 days after vaccination | ≥ 14 days after vaccination
  Number of participants experiencing RSV-LRTD (RSV B) ≥ 14 days after vaccination
Presence of the first episode of RSV-LRTD (RSV A and/or RSV B and by each one) by age group | ≥ 14 days after vaccination
  Number of participants experiencing RSV-LRTD (RSV A and/or B and by each one) by age group
Presence of the first episode of RSV LRTD (RSV A and/or RSV B and by each one) by baseline comorbidities | ≥ 14 days after vaccination
  Number of participants experiencing RSV-LRTD (RSV A and/or B and by each one) by baseline comorbidities
Presence of the first episode of RSV LRTD (RSV A and/or RSV B and by each one) by baseline frailty status | ≥ 14 days after vaccination
  Number of participants experiencing RSV-LRTD (RSV A and/or B and by each one) by baseline frailty status
Presence of hospitalization due to RSV-ARD and/or RSV-LRTD | ≥ 14 days after vaccination
  Number of participants hospitalized due to RSV-ARD and/or RSV-LRTD
Duration (number of days) of RSV LRTD episodes (RSV A and/or RSV B) | ≥ 14 days after vaccination
  Duration (number of days) of RSV LRTD episodes (RSV A and/or RSV B)
Duration (number of days) of RSV ARD episodes (RSV A and/or RSV B) | ≥ 14 days after vaccination
  Duration (number of days) of RSV ARD episodes (RSV A and/or RSV B)
Presence of the first episode of severe RSV LRTD (RSV A and/or RSV B and by each one) occurring ≥ 14 days after vaccination | ≥ 14 days after vaccination
  Number of participants experiencing severe RSV-LRTD (RSV A and/or B and by each one)
RSV A serum neutralizing antibodies (nAb) titers at pre vaccination (D01) and 28 days (D29) post vaccination in the Immunogenicity Subset | Day 1 and Day 29
  RSV A serum neutralizing antibodies (nAb) titers at pre vaccination (D01) and 28 days (D29) post vaccination in the Immunogenicity Subset
RSV B serum nAb titers at pre vaccination (D01) and 28 days (D29) post vaccination in the Immunogenicity Subset | Day 1 and Day 29
  RSV B serum nAb titers at pre vaccination (D01) and 28 days (D29) post vaccination in the Immunogenicity Subset
Serum anti-F immunoglobulin G (IgG) antibody (Ab) titers at pre-vaccination (D01) and 28 days (D29) post vaccination in the Immunogenicity Subset | Day 1 and Day 29
  Serum anti-F immunoglobulin G (IgG) antibody (Ab) titers at pre-vaccination (D01) and 28 days (D29) post vaccination in the Immunogenicity Subset
RSV A serum nAb titers at 6 months post-vaccination in the Immunogenicity Subset | Month 6
  RSV A serum nAb titers at 6 months post-vaccination in the Immunogenicity Subset
RSV B serum nAb titers at 6 months post-vaccination in the Immunogenicity Subset | Month 6
  RSV B serum nAb titers at 6 months post-vaccination in the Immunogenicity Subset
Serum anti-F IgG Ab titers at 6 months post-vaccination in the Immunogenicity Subset | Month 6
  Serum anti-F IgG Ab titers at 6 months post-vaccination in the Immunogenicity Subset
Presence of solicited injection site or systemic reactions | Within 7 days after primary vaccination
  Number of participants reporting:
  * injection site reactions: pain, erythema and swelling
  * systemic reactions: fever, headache, fatigue, myalgia, arthralgia and chills
Presence of unsolicited immediate systemic adverse events (AEs) | Within 30 minutes after primary vaccination
  Number of participants experiencing an unsolicited immediate systemic adverse event
Presence of unsolicited AEs | Within 28 days after primary vaccination
  Number of participants experiencing unsolicited AEs
Presence of serious adverse events (SAEs) | Throughout study (approximately 6 months)
  Number of participants experiencing SAEs
Presence of medically attended adverse events (MAAEs) | Throughout study (approximately 6 months)
  Number of participants experiencing MAAEs
Presence of adverse events of special interest (AESIs) | Throughout study (approximately 6 months)
  Number of participants experiencing AESIs

CONTACTS AND LOCATIONS:
Locations (25):
- Australia (5):
  - Investigational Site Number : 0360003, Botany, New South Wales
  - Investigational Site Number : 0360004, Sippy Downs, Queensland
  - Investigational Site Number : 0360001, Southport, Queensland
  - Investigational Site Number : 0360002, Camberwell, Victoria
  - Investigational Site Number : 0360005, Norwood
- Chile (6):
  - Investigational Site Number : 1520005, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520001, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520004, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520006, Concepción, Región del Biobío
  - Investigational Site Number : 1520002, Santiago
  - Investigational Site Number : 1520008, Santiago
- Colombia (7):
  - Investigational Site Number : 1700004, Aguazul
  - Investigational Site Number : 1700002, Barranquilla
  - Investigational Site Number : 1700006, Bogotá
  - Investigational Site Number : 1700007, Cali
  - Investigational Site Number : 1700003, Girardot
  - Investigational Site Number : 1700005, Ibagué
  - Investigational Site Number : 1700001, Quindío
- Dominican Republic (2):
  - Investigational Site Number : 2140001, Santo Domingo
  - Investigational Site Number : 2140002, Santo Domingo
- Honduras (3):
  - Investigational Site Number : 3400001, San Pedro Sula
  - Investigational Site Number : 3400003, Tegucigalpa
  - Investigational Site Number : 3400002, Tegucugalpa
- Mexico (2):
  - Investigational Site Number : 4840002, León, Guanajuato
  - Investigational Site Number : 4840003, Querétaro

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org